CLINICAL TRIAL: NCT01722097
Title: Recovery After Laparoscopic Hysterectomy With Deep Neuromuscular Blockade and Low Intra-abdominal Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Matias Vested Madsen, research assistent, MD, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMBDK2012; 2012-003787-51 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Neuromuscular Blockade; Pain; Laparoscopy
MeSH Terms: conditions — Pain | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep neuromuscular blockade (Active Comparator): Drug: Rocuronium Intravenous use: 0.3 mg/kg before intubation and 0,7 mg after intubation followed by infusion with 0,3-0,4 mg/kg/h Other Name: Esmeron
  Interventions: Drug: Rocuronium
- Moderate neuromuscular blockade (Placebo Comparator): Drug: Rocuronium Intravenous use: 0,3 mg/kg followed by NaCl-infusion Other Name: Esmeron
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rocuronium
  Arms: Deep neuromuscular blockade
Drug: placebo
  Arms: Moderate neuromuscular blockade

SUMMARY:
The purpose of this study on laparoscopic hysterectomy is to investigate postoperative pain. Patients are allocated to either deep neuromuscular blockade and low intra-abdominal pressure (8 mmHg) or moderate neuromuscular blockade and usual intra-abdominal pressure (12 mmHg).

Primary hypothesis:

Deep neuromuscular blockade and low intra-abdominal pressure (8 mmHg) reduces postoperative pain compared to moderate neuromuscular blockade and intra-abdominal pressure (12 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic hysterectomy (total/subtotal)
* Can read and understand Danish
* Informed consent

Exclusion Criteria:

* BMI > 30 kg/cm2
* Known allergy to medications that are included in the project
* Severe renal disease, defined by S-creatinine > 0,200 mmol/L, GFR < 30ml/min or hemodialysis)
* Neuromuscular disease that may interfere with neuromuscular data
* Lactating
* Impaired liver function
* Indication for rapid sequence induction (esophageal reflux/ hiatus hernia/other cause)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Gätke, MD, ph.d., Study Chair — Department of anesthesia, Herlev Hospital; Matias Vested Maden, MD, Principal Investigator — Department of anesthesia, Herlev Hospital
Locations (1):
- Department of anesthesia and department of minimal invasive gynecology, Aleris-Hamlet, Søborg, Denmark

REFERENCES:
- [Derived] Madsen MV, Istre O, Springborg HH, Staehr-Rye AK, Rosenberg J, Lund J, Gatke MR. Deep neuromuscular blockade and low insufflation pressure during laparoscopic hysterectomy. Dan Med J. 2017 May;64(5):A5364. PMID 28552090
- [Derived] Madsen MV, Istre O, Staehr-Rye AK, Springborg HH, Rosenberg J, Lund J, Gatke MR. Postoperative shoulder pain after laparoscopic hysterectomy with deep neuromuscular blockade and low-pressure pneumoperitoneum: A randomised controlled trial. Eur J Anaesthesiol. 2016 May;33(5):341-7. doi: 10.1097/EJA.0000000000000360. PMID 26479510

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Neuromuscular Blockade: Drug: Rocuronium Intravenous use: 0.3 mg/kg before intubation and 0,7 mg after intubation followed by infusion with 0,3-0,4 mg/kg/h Other Name: Esmeron
  Rocuronium
- Moderate Neuromuscular Blockade: Drug: Rocuronium Intravenous use: 0,3 mg/kg followed by NaCl-infusion Other Name: Esmeron
  placebo
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Started | 55 | 55
Completed | 49 | 50
Not Completed | 6 | 5
Not completed — Patient sheets not returned | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (5) | 48 (5) | 47 (5)
Sex/Gender, Customized [Number; unit: participants] — In total 110 women participated in the study
  participants
    women | 55 | 55 | 110
Region of Enrollment [Number; unit: participants]
  Denmark | 55 | 55 | 110
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (3.0) | 24.2 (3.1) | 23.6 (3.1)
American Society of Anesthesiologists Physical Status Classification 1 [Number; unit: participants] — American Society of Anesthesiologists (ASA) PHYSICAL STATUS CLASSIFICATION SYSTEM 1-6.
  1. A normal healthy patient
  2. A patient with mild systemic disease
  3. A patient with severe systemic disease
  4. A patient with severe systemic disease that is a constant threat to life
  5. A moribund patient who is not expected to survive without the operation
  6. A declared brain-dead patient whose organs are being removed for donor purposes
  participants | 52 | 49 | 101
Parity (full term pregnancies) [Median (Full Range); unit: pregnancies] | 2 [0 to 4] | 2 [0 to 4] | 2 [0 to 4]
Previous abdominal surgery [Number; unit: participants] | 26 | 35 | 61
Subtotal hysterectomy [Number; unit: participants] | 26 | 27 | 53
American Society of Anesthesiologists Physical Status Classification 2 [Number; unit: participants] | 3 | 6 | 9
Total hysterectomy [Number; unit: participants] | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Pain
Description: Number of participants with shoulder pain or discomfort (VAS > 20) in the shoulder region within 14 days after operation.
  VAS 0-100: Visual analouge scale for assessment of pain ranging from no pain (value 0) to worst kind of pain (value 100).
Time Frame: within 14 days
Measure: Number; unit: participants
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Number analyzed (Participants) | 49 | 50
participants | 14 | 30

2. Secondary Outcome: Pain (Assessed on a 0-100 Visual Analouge Scale (VAS): 0 no Pain, 100 Worst Kind of Pain)
Description: Pain (shoulder-, incisional-, abdominal - and overall pain) estimated as area under the curve (AUC) from 0 till 4 days after operation.
  Pain (shoulder-, incisional-, abdominal - and overall pain) estimated as area under the curve (AUC) from 0 till 14 days after operation.
  Pain was assessed: preoperatively, at arrival to the postanesthesia care unit, 2 hours after surgery, 4 hours after surgery, 8 hours after surgery, at discharge from hospital, and once daily at day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14 after surgery.
Time Frame: within 14 days
Measure: Median (Inter-Quartile Range); unit: units on a scale*days
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Number analyzed (Participants) | 49 | 50
units on a scale*days
  VAS shoulder pain 4 days AUC | 16.4 [5.8 to 44.7] | 28.5 [6.3 to 52.2]
  VAS shoulder pain 14 days AUC | 27.6 [8.2 to 67.9] | 36.3 [9.7 to 86.6]
  VAS incisional pain 4 days AUC | 88.4 [33.8 to 189.3] | 102.2 [35.8 to 159.1]
  VAS incisional pain 14 days AUC | 144.6 [62.0 to 291.6] | 150.8 [56.8 to 306.3]
  VAS abdominal pain 4 days AUC | 102.4 [50.0 to 213.2] | 114.1 [57.8 to 207.5]
  VAS abdominal pain 14 days AUC | 190.8 [103.2 to 366.8] | 215.5 [109.5 to 396.3]
  VAS overall pain 4 days AUC | 101.7 [51.9 to 200.8] | 129.8 [79.0 to 198.1]
  VAS overall pain 14 days AUC | 190.2 [118.9 to 402.5] | 256.9 [121.3 to 403.7]

3. Other Pre Specified Outcome: Patient-movements
Description: Number of unintended and unwanted patient-movements registered by the surgeon
Time Frame: During surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Deep Neuromuscular Blockade | Moderate Neuromuscular Blockade
Serious Adverse Events (participants affected / at risk) | 4/55 | 3/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Neuromuscular Blockade (N=55) | Moderate Neuromuscular Blockade (N=55)
Infection after surgery (Infections and infestations) | 2 (2) | 1 (1)
Lesion of the bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Vesicovaginal fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Postoperative bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)
hematoma (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes